CLINICAL TRIAL: NCT04063293
Title: The Effect of Platelet Rich Plasma Injection Into the Anal Sphincters on Fecal Incontinence and Quality of Life in Incontinent Patients Had Treated With Low Anterior Resection for Rectal Cancer
Brief Title: PRP Injection Into Anal Sphincters for Fecal Incontinence
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMU260702
Record Dates: First submitted 2019-08-15; First posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Fecal Incontinence
Keywords: fecal incontinence; platelet rich plasma; PRP; injection
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Intervention Model Description: The injection will be performed in operation room under general anesthesia with either IV sedation of laryngeal mask airway (LMA) sedation. In case a perfect relaxation will not be achieved, then the patient will be intubated. The patient will be positioned as gynecological position. 10 cc of PRP will be directly injected in external muscles at 8 locations under the guidance of endoanal ultrasound. The final condition of the sphincters will be pictured with the device. The same surgeon (MCH) will perform all procedures. No antibiotics will be used. Local anesthetics will not be injected. If the patient will feel pain after the operation, he/she will be free to use oral painkillers. The patient will be discharged from the hospital on the same night or the day after according to the patient's desire. Patients will be questioned for possible PRP complications during the hospitalization period, and they will be asked to report anytime during the study period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRP injection (Experimental): PRP is prepared using a special device (VS-400, Genesis Comp, Korea). For each application a kit (e+ PRP, Genesis Comp, Korea) will be used. 18 cc of venous blood will be collected from the patient into the syringe with 2 cc of anticoagulant, and will be gently inverted. The sample will be slowly injected into the e+ PRP kit. The kit will be centrifuged under 1,500G for 4 minutes, which will separate the blood components into 3 different layers. The rot at the top of the kit will be pressed until the bottom of the piston will touch the red blood cell layer, and the rot will be turned clockwise to close it. The cap will be opened and the small syringe will be connected to the cap for extracting PRP. The injection will be performed in operation room under general anesthesia with either IV sedation of laryngeal mask airway (LMA) sedation. 10 cc of PRP will be directly injected in external muscles at 8 locations under the guidance of endoanal ultrasound
  Interventions: Biological: Platelet Rich Plasma

INTERVENTIONS:
Biological: Platelet Rich Plasma — PRP injection into tha anal canal in patients underwent low anterior resection for rectal cancer
  Other Names: PRP

SUMMARY:
The treatment of fecal incontinence after low anterior resection is problematic, and not always able to increase quality of life. Biofeedback and rehabilitation therapies are harmless and easy to use; thus, generally selected as the initial treatment modalities, however may be effective in a small portion of patients. More complex treatment techniques including sacral nerve stimulation decrease the severity of symptoms, however the implantation of the device is a costly, staged procedure. Little is known about the effectiveness of other techniques such as injectable substances on incontinence observed after low anterior resection. There is no study evaluating the safety and effectiveness of platelet rich plasma (PRP) injection for incontinent patients after low anterior resection.

DETAILED DESCRIPTION:
Rectal cancer is a common problem worldwide and the standard potentially curative treatment for locally advanced disease includes radical surgery appreciating oncological principals. Sphincter-saving procedures have been practiced in order to prevent a permanent stoma; however, patients underwent low anterior resection may suffer from several problems including incontinence particularly if the initial tumor is located too close to the anal canal. The actual frequency of incontinence is still unknown because of wide variation rates in several reports ranging between 0 to 80%; and may be a long-term problem since a series has presented an incidence of 36% 10 years after surgery.

Several mechanisms may cause incontinence after low anterior resection, thus several therapeutic instruments have been described considering the underlying reason. The most reasonable suspect is probably an injury to the sphincters at the time of surgery or secondary to preoperative radiation therapy, which is a commonly used modality in order to reduce local recurrence and increase the possibility of sphincter-saving procedures with the shrinkage of the tumor. Surgery and/or (chemo)radiation may not only generate sphincter injury, but also cause nerve damage and consequent denervation of the sphincters. Internal sphincters are responsible for resting pressure. Incontinence is more often and obvious if an intersphincteric resection with a hand-sewn coloanal anastomosis is attempted, since this procedure indicates the removal of internal sphincters. Several studies have revealed that up to 20% of patients have internal sphincter injuries after low anterior resection proven with endoanal ultrasound or manometer; and diminution in size of sphincters and decrease in resting pressure are correlated with incontinence grade. Mechanical anal sphincter injury may occur during the insertion of stapler; thus, incontinence may also be observed in patients with more proximally located tumors. The effect of radiation therapy on sphincter functions is also well-known, and a prospective randomized trial has shown that radiotherapy is significantly increasing incontinence rate. Another mechanism in incontinence may be related to the reduction of the capacity of neorectum, since descending colon, which is the reconstructing organ in most cases is narrower than rectum itself. Several reservoir techniques including coloplasty, colonic j-pouch and side-to-end anastomosis have been described in order to increase pooling volume of neorectum. Some other factors including decrease in sensitivity of anal canal and anal transitional zone, alteration in rectoanal inhibitory reflex, motility dysfunction of neorectum and incomplete evacuation may separately cause incontinence or increase the severity of symptoms. Instead of a sole origin, a combination of several reasons may be present at the same time making the problem more complex and the solution tougher. The treatment of incontinence is problematic, and not always able to increase quality of life. Biofeedback and rehabilitation therapies are harmless and easy to use; thus, generally selected as the initial treatment modalities, however may be effective in a small portion of patients. More complex treatment techniques including sacral nerve stimulation decrease the severity of symptoms, however the implantation of the device is a costly, staged procedure. Little is known about the effectiveness of other techniques such as injectable substances on incontinence observed after low anterior resection. Some patients may require fecal diversion in order to achieve a better quality of life.

Platelet Rich Plasma (PRP) is a thrombocyte enriched liquid, and it increases cell proliferation and collagen formation where it is injected. Platelets activate some growth factors, cytokines and other bioactive mediators, and consequently initiate and regulate wound-healing period. PRP has been used in several chronic diseases for initiating and fastening the reconstruction phase, particularly for the tendon, muscle, ligament and articular system related injuries and inflammatory situations. The effects of PRP on symptoms and healing rate in patients with lateral epicondylitis and its superiority over bupivacaine or steroid injections have been shown in cohort and prospective randomized trials. PRP is also tested for the treatment of perianal fistula. When PRP injection is combined with mucosal advancement flap procedure, it has been shown to decrease the recurrence rate. In an animal model, PRP injection into the gastrocnemius muscle has shown to increase the strength of the muscle healing. Although it has a potential, -to the best to our knowledge- there is no study evaluating the safety and effectiveness of PRP injection for incontinent patients after low anterior resection.

Methods:

This project is a single arm, cohort study evaluating the safety and effectiveness of PRP injection into the anal sphincter on incontinence and related quality of life in incontinent patients after low anterior resection for rectal cancer. All participating patients will be informed about the protocol and PRP application, and informed consent will be obtained. The study will be run at Department of General Surgery at Istanbul Medipol University Medical School (IMU) and be completed in 24 months. Local Ethical Committee has approved the protocol (protocol number: 66291034-29) and The Scientific and Technological Research Council of Turkey (TUBITAK) has granted the study (project number: 117s133). First patient accrual is planned to happen before August 2019. For the first year, only the patients who had their previous cancer operation at IMU will be included to the study, but in case of a shortage in number of patients by the end of August 2020, the inclusion of the patients who had their initial surgeries in other institutions will be permitted.

Local Ethical Committee and governors of TUBITAK will be free to monitor the trial progress at any time. Actual status of the study will be reported to TUBITAK for observation and for the continuity of grant imbursements annually (twice during the study period) and after the finalization of data analysis and publishing. Interim analysis will not be stated, since the design has not been classified as high risk.

ELIGIBILITY:
Inclusion Criteria:

* incontinent patients after low anterior resection for rectal cancer

Exclusion Criteria:

* There are 2 types of exclusion criteria

A. Patients who will not be suitable for initial tests:

1. Patients younger than 18 or older than 80
2. Pregnant or lactating women
3. Patients received pelvic radiation after the initial cancer surgery
4. Patients with local recurrence
5. Patients with irresectable metastasis (patients with resectable liver and/or lung metastasis will be included after metastasectomy, but patients with peritoneal metastasis who will be candidate for peritonectomy will not be included)
6. Patients under chemotherapy
7. Patients confess incontinence prior to initial cancer surgery
8. Contraindication for PRP injection: active infection, thrombocytopenia, anemia (Hgb <10 gr/dl), allergy for buffalo thrombin
9. If the interval after the final surgery less than 12 months
10. Patient refusal

B. Patients who will be excluded according to manometer and/or endoanal ultrasound findings. Only the patients with an acceptable volume of healthy anal sphincters, an adequate reservoir capacity of neorectum and decreased sphincter strength will be included to the study after ruling out a full-thickness external sphincter tear will be the subjects of the evaluation. These patients will be excluded prior to PRP injection:

1. If manometer reveals normal resting (59-74 mm) and squeeze (124-152 mm) pressure (No clue for decreased sphincter strength)
2. If manometer reveals higher than normal volume (17-23 cc) for the first sensation, since it shows reduction of rectal sensitivity
3. If manometer reveals lessened maximum tolerable volume (MTV), since the continence may be related to the reduced volume of neorectum (For healthy volunteers the normal level of MTV is between 216 cc and 266 cc. Although normal level for neorectum after low anterior resection is not known, in a study it is accepted to be more than 60 cc as the current study [28]).
4. No or minimal external sphincter volume during: for inclusion the length, wide and volume of the external sphincter should be at least 16.1 mm, 6.8 mm and 6.3 cc, respectively (for inclusion all 3 measures should fulfilled). Although the actual minimal volume of external sphincter preventing incontinence is not indicated, in this study the minimal volume in healthy volunteers has been accepted [29,30].
5. Endoanal ultrasound examination revealing full-thickness tear in external sphincter.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-08-15 (Estimated); Study Completion 2021-02-15 (Estimated)

PRIMARY OUTCOMES:
Wexner fecal incontinence score change | baseline and 6 months after PRP injection
  This scoring system cross-tabulates frequencies and different anal incontinence presentations (Gas/Liquid/Solid/Pad use/Need for lifestyle alterations) and sums the returned score to a total of 0-20 (where 0 = perfect continence and 20 = complete incontinence). Each of the incontinence presentations is graded equally.

SECONDARY OUTCOMES:
St Mark's (Vaizey) score | baseline and 6 months after PRP injection
  analyzes different incontinence situations (solid, liquid, gas) and frequencies. Lifestyle alteration, need to wear a pad, taking constipating medicaiton and Lack of ability to defer defecation for 15 minutes. Minimum score is 0 = perfect continence; maximum score is 24 = totally incontinent.
Pescatori incontinence score | baseline and 6 months after PRP injection
  The Pescatori AI score is a grading system that combines both degree of incontinence (flatus-mucus/liquid stool/solid stool) with frequency. Incontinence ratings of A, B and C indicate AI for flatus/mucus, liquid stool, and solid stool, respectively; frequency scores of 1, 2 and 3 indicate occasional, weekly, and daily AI. A score of zero is given for normal continence. The combined score is the sum of the degree and the frequency. The minimum score is 0 and the maximum score is 6
Fecal Incontinence Quality of Life Questionnaires | baseline and 6 months after PRP injection
  a disease-specific tool, was designed to evaluate the impact of FI on four aspects of patients' QOL: lifestyle; coping behavior; depression or self perception; and level of embarrassment. The scale is composed of a total of 29 items; these items form four scales: Lifestyle (10 items), Coping/Behavior (9 items), Depression/Self-Perception (7 items), and Embarrassment (3 items).Each aspect is described as a score measured on a scale between 1 and 4, where 1 is very affected and 4 is not affected
SF-36 Questionnairy | baseline and 6 months after PRP injection
  The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100 Lower scores = more disability, higher scores = less disability Sections: Vitality, Physical functioning, Bodily pain, General health perceptions, Physical role functioning, Emotional role functioning, Social role functioning, Mental health
Anal resting pressure | baseline and 6 months after PRP injection
Maximal squeeze pressure | baseline and 6 months after PRP injection
Isolated squeeze pressure | baseline and 6 months after PRP injection
Initial sensation volume | baseline and 6 months after PRP injection
Volume for defecation need | baseline and 6 months after PRP injection
Maximal tolerable volume | baseline and 6 months after PRP injection
Number of participants with PRP injection-related adverse events as assessed by CTCAE v4.0 | up to 6 months after PRP injection
  PRP injection safety

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa C Haksal, MD, Principal Investigator — Istanbul Medipol University Medical School; Mustafa Oncel, Prof, Study Chair — Istanbul Medipol University Medical School
Locations (1):
- Istanbul Medipol University Medical School, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: after the final date of the study, for 1 year
Access Criteria: related data will be shared with interested clinicians to use the info in their studies and to re-analyse our findings. Contact will be via e-mail of the PI

REFERENCES:
- [Background] Ziv Y, Zbar A, Bar-Shavit Y, Igov I. Low anterior resection syndrome (LARS): cause and effect and reconstructive considerations. Tech Coloproctol. 2013 Apr;17(2):151-62. doi: 10.1007/s10151-012-0909-3. Epub 2012 Oct 18. PMID 23076289
- [Background] Bryant CL, Lunniss PJ, Knowles CH, Thaha MA, Chan CL. Anterior resection syndrome. Lancet Oncol. 2012 Sep;13(9):e403-8. doi: 10.1016/S1470-2045(12)70236-X. PMID 22935240
- [Background] Peeters KC, van de Velde CJ, Leer JW, Martijn H, Junggeburt JM, Kranenbarg EK, Steup WH, Wiggers T, Rutten HJ, Marijnen CA. Late side effects of short-course preoperative radiotherapy combined with total mesorectal excision for rectal cancer: increased bowel dysfunction in irradiated patients--a Dutch colorectal cancer group study. J Clin Oncol. 2005 Sep 1;23(25):6199-206. doi: 10.1200/JCO.2005.14.779. PMID 16135487
- [Background] Lundby L, Krogh K, Jensen VJ, Gandrup P, Qvist N, Overgaard J, Laurberg S. Long-term anorectal dysfunction after postoperative radiotherapy for rectal cancer. Dis Colon Rectum. 2005 Jul;48(7):1343-9; discussion 1349-52; author reply 1352. doi: 10.1007/s10350-005-0049-1. PMID 15933797
- [Background] Ridolfi TJ, Berger N, Ludwig KA. Low Anterior Resection Syndrome: Current Management and Future Directions. Clin Colon Rectal Surg. 2016 Sep;29(3):239-45. doi: 10.1055/s-0036-1584500. PMID 27582649
- [Background] Ishiyama G, Hinata N, Kinugasa Y, Murakami G, Fujimiya M. Nerves supplying the internal anal sphincter: an immunohistochemical study using donated elderly cadavers. Surg Radiol Anat. 2014 Dec;36(10):1033-42. doi: 10.1007/s00276-014-1289-3. Epub 2014 Apr 2. PMID 24691518
- [Background] Konanz J, Herrle F, Weiss C, Post S, Kienle P. Quality of life of patients after low anterior, intersphincteric, and abdominoperineal resection for rectal cancer--a matched-pair analysis. Int J Colorectal Dis. 2013 May;28(5):679-88. doi: 10.1007/s00384-013-1683-z. Epub 2013 Apr 10. PMID 23571868
- [Background] Farouk R, Duthie GS, Lee PW, Monson JR. Endosonographic evidence of injury to the internal anal sphincter after low anterior resection: long-term follow-up. Dis Colon Rectum. 1998 Jul;41(7):888-91. doi: 10.1007/BF02235373. PMID 9678375
- [Background] Hirano A, Koda K, Kosugi C, Yamazaki M, Yasuda H. Damage to anal sphincter/levator ani muscles caused by operative procedure in anal sphincter-preserving operation for rectal cancer. Am J Surg. 2011 Apr;201(4):508-13. doi: 10.1016/j.amjsurg.2009.12.016. Epub 2010 Sep 29. PMID 20883975
- [Background] Ho YH, Tsang C, Tang CL, Nyam D, Eu KW, Seow-Choen F. Anal sphincter injuries from stapling instruments introduced transanally: randomized, controlled study with endoanal ultrasound and anorectal manometry. Dis Colon Rectum. 2000 Feb;43(2):169-73. doi: 10.1007/BF02236976. PMID 10696889
- [Background] Tomita R, Igarashi S, Fujisaki S. Studies on anal canal sensitivity in patients with or without soiling after low anterior resection for lower rectal cancer. Hepatogastroenterology. 2008 Jul-Aug;55(85):1311-4. PMID 18795679
- [Background] Kim KH, Yu CS, Yoon YS, Yoon SN, Lim SB, Kim JC. Effectiveness of biofeedback therapy in the treatment of anterior resection syndrome after rectal cancer surgery. Dis Colon Rectum. 2011 Sep;54(9):1107-13. doi: 10.1097/DCR.0b013e318221a934. PMID 21825890
- [Background] Visser WS, Te Riele WW, Boerma D, van Ramshorst B, van Westreenen HL. Pelvic floor rehabilitation to improve functional outcome after a low anterior resection: a systematic review. Ann Coloproctol. 2014 Jun;30(3):109-14. doi: 10.3393/ac.2014.30.3.109. Epub 2014 Jun 23. PMID 24999460
- [Background] Tan E, Ngo NT, Darzi A, Shenouda M, Tekkis PP. Meta-analysis: sacral nerve stimulation versus conservative therapy in the treatment of faecal incontinence. Int J Colorectal Dis. 2011 Mar;26(3):275-94. doi: 10.1007/s00384-010-1119-y. Epub 2011 Jan 29. PMID 21279370
- [Background] Schwandner O. Sacral neuromodulation for fecal incontinence and "low anterior resection syndrome" following neoadjuvant therapy for rectal cancer. Int J Colorectal Dis. 2013 May;28(5):665-9. doi: 10.1007/s00384-013-1687-8. Epub 2013 Apr 5. PMID 23559414
- [Background] Soerensen MM, Lundby L, Buntzen S, Laurberg S. Intersphincteric injected silicone biomaterial implants: a treatment for faecal incontinence. Colorectal Dis. 2009 Jan;11(1):73-6. doi: 10.1111/j.1463-1318.2008.01544.x. Epub 2008 Apr 28. PMID 18462216
- [Background] Kim DW, Yoon HM, Park JS, Kim YH, Kang SB. Radiofrequency energy delivery to the anal canal: is it a promising new approach to the treatment of fecal incontinence? Am J Surg. 2009 Jan;197(1):14-8. doi: 10.1016/j.amjsurg.2007.11.023. Epub 2008 Jul 9. PMID 18614149
- [Background] Foster TE, Puskas BL, Mandelbaum BR, Gerhardt MB, Rodeo SA. Platelet-rich plasma: from basic science to clinical applications. Am J Sports Med. 2009 Nov;37(11):2259-72. doi: 10.1177/0363546509349921. PMID 19875361
- [Background] Mishra A, Pavelko T. Treatment of chronic elbow tendinosis with buffered platelet-rich plasma. Am J Sports Med. 2006 Nov;34(11):1774-8. doi: 10.1177/0363546506288850. Epub 2006 May 30. PMID 16735582
- [Background] Peerbooms JC, Sluimer J, Bruijn DJ, Gosens T. Positive effect of an autologous platelet concentrate in lateral epicondylitis in a double-blind randomized controlled trial: platelet-rich plasma versus corticosteroid injection with a 1-year follow-up. Am J Sports Med. 2010 Feb;38(2):255-62. doi: 10.1177/0363546509355445. PMID 20448192
- [Background] Gosens T, Peerbooms JC, van Laar W, den Oudsten BL. Ongoing positive effect of platelet-rich plasma versus corticosteroid injection in lateral epicondylitis: a double-blind randomized controlled trial with 2-year follow-up. Am J Sports Med. 2011 Jun;39(6):1200-8. doi: 10.1177/0363546510397173. Epub 2011 Mar 21. PMID 21422467
- [Background] Gottgens KW, Vening W, van der Hagen SJ, van Gemert WG, Smeets RR, Stassen LP, Baeten CG, Breukink SO. Long-term results of mucosal advancement flap combined with platelet-rich plasma for high cryptoglandular perianal fistulas. Dis Colon Rectum. 2014 Feb;57(2):223-7. doi: 10.1097/DCR.0000000000000023. PMID 24401885
- [Background] Moreno-Serrano A, Garcia-Diaz JJ, Ferrer-Marquez M, Alarcon-Rodriguez R, Alvarez-Garcia A, Reina-Duarte A. Using autologous platelet-rich plasma for the treatment of complex fistulas. Rev Esp Enferm Dig. 2016 Mar;108(3):123-8. doi: 10.17235/reed.2016.3946/2015. PMID 26856400
- [Background] Pinheiro CL, Peixinho CC, Esposito CC, Manso JE, Machado JC. Ultrasound biomicroscopy and claudication test for in vivo follow-up of muscle repair enhancement based on platelet-rich plasma therapy in a rat model of gastrocnemius laceration. Acta Cir Bras. 2016 Feb;31(2):103-10. doi: 10.1590/S0102-865020160020000004. PMID 26959619
- [Background] Cong JC, Chen CS, Ma MX, Xia ZX, Liu DS, Zhang FY. Laparoscopic intersphincteric resection for low rectal cancer: comparison of stapled and manual coloanal anastomosis. Colorectal Dis. 2014 May;16(5):353-8. doi: 10.1111/codi.12573. PMID 24460588
- [Background] Hong KD, Kim JS, Ji WB, Um JW. Midterm outcomes of injectable bulking agents for fecal incontinence: a systematic review and meta-analysis. Tech Coloproctol. 2017 Mar;21(3):203-210. doi: 10.1007/s10151-017-1593-0. Epub 2017 Mar 1. PMID 28251356
- [Background] Felt-Bersma RJ, Sloots CE, Poen AC, Cuesta MA, Meuwissen SG. Rectal compliance as a routine measurement: extreme volumes have direct clinical impact and normal volumes exclude rectum as a problem. Dis Colon Rectum. 2000 Dec;43(12):1732-8. doi: 10.1007/BF02236859. PMID 11156459
- [Background] Olsen IP, Augensen K, Wilsgaard T, Kiserud T. Three-dimensional endoanal ultrasound assessment of the anal sphincters during rest and squeeze. Acta Obstet Gynecol Scand. 2008;87(6):669-74. doi: 10.1080/00016340802088346. PMID 18568467
- [Background] Gregory WT, Boyles SH, Simmons K, Corcoran A, Clark AL. External anal sphincter volume measurements using 3-dimensional endoanal ultrasound. Am J Obstet Gynecol. 2006 May;194(5):1243-8. doi: 10.1016/j.ajog.2005.10.822. Epub 2006 Apr 21. PMID 16647906
- [Background] Vaizey CJ, Carapeti E, Cahill JA, Kamm MA. Prospective comparison of faecal incontinence grading systems. Gut. 1999 Jan;44(1):77-80. doi: 10.1136/gut.44.1.77. PMID 9862829
- [Background] Rullier E, Laurent C, Bretagnol F, Rullier A, Vendrely V, Zerbib F. Sphincter-saving resection for all rectal carcinomas: the end of the 2-cm distal rule. Ann Surg. 2005 Mar;241(3):465-9. doi: 10.1097/01.sla.0000154551.06768.e1. PMID 15729069